CLINICAL TRIAL: NCT00840983
Title: Effects of Delayed Cord Clamping in Very Low Birth Weight (VLBW) Infants
Brief Title: Effects of Delayed Cord Clamping in Very Low Birth Weight Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Judith S Mercer, Professor Emerita, University of Rhode Island
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Mercer-K23-03; R01NR010015-01A2 (NIH)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Bronchopulmonary Dysplasia; Necrotizing Enterocolitis; Intraventricular Hemorrhage; Late Onset Neonatal Sepsis; Motor Skills Disorders
Keywords: delayed cord clamping; very low birthweight infant; bronchopulmonary dysplasia; intraventricular hemorrhage; motor function
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Enterocolitis, Necrotizing; Neonatal Sepsis; Motor Skills Disorders | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-Immediate Cord Clamping (No Intervention): infants received the routine care of immediate clamping of the umbilical cord
- 2-Delayed Cord Clamping (Experimental): after birth, cord clamping was delayed 30 to 45 seconds while infant was held lower than the level of the placenta.
  Interventions: Procedure: delayed cord clamping

INTERVENTIONS:
Procedure: delayed cord clamping — cord clamping was delayed for 30 to 45 seconds and infant was held lower than the level of the placenta
  Other Names: cord clamping time
  Arms: 2-Delayed Cord Clamping

SUMMARY:
The purpose of this study was to see if a brief delay in cord clamping for 30 to 45 seconds would result in higher hematocrit levels, fewer transfusions, healthier lungs, and better motor function at 40 wks and 7 months of age.

DETAILED DESCRIPTION:
When cord clamping is delayed at birth or the cord is milked, infants receive a placental transfusion of 10-15 mL/kg during the first few minutes of life. This additional blood improves hemodynamic stability and may reduce the risk of intraventricular hemorrhage (IVH) and the vulnerability of infants to inflammatory processes. This blood also contains stem cells that are important in repairing tissue and building immunocompetence.

The current randomized controlled trial prospectively tested the effects of DCC for 30-45 seconds followed by 1 cord milking with the aim of confirming our prior work and providing long-term follow-up. Our a priori hypotheses were that DCC would reduce the incidence of IVH, LOS, and result in better motor function at 18-22 months.

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant with gestation 24 to 31.6 weeks of singleton pregnancy by obstetrical evaluation
* Obstetrician's approval of enrollment into study
* Parental consent
* Any mode of birth will be included

Exclusion Criteria:

* Obstetrician's refusal to enroll infants
* Parental refusal for consent
* Prenatally-diagnosed major congenital anomalies [or multiple gestations]
* Intent to withhold or withdraw care
* Severe or multiple maternal illnesses, frank vaginal bleeding, placenta abruption or previa
* Mothers who are institutionalized or psychotic

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-08; Primary Completion 2005-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
VLBW infants in the delayed clamped group will have less chronic lung disease at 36 weeks postmenstrual age compared to VLBW infants in the immediate cord clamped grouped | 36 wks postmenstrual age
VLBW infants in the delayed clamped group will have fewer incidences of suspected necrotizing enterocolitis during the NICU stay when compared with VLBW infants in the immediate cord clamped group | Hospital discharge
VLBW infants in the delayed clamped group will have better motor function by 6 to corrected age when compared with VLBW infants in the immediate cord clamped group | 7 months corrected age

SECONDARY OUTCOMES:
Infants in the delayed cord clamping group will have less IVH than infants in the immediate clamping group | NICU stay
Infants in the delayed clamping group will hvae less late onset sepsis than infants in the immediate clamping group. | NICU Stay

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Mercer, PhD, CNM, Principal Investigator — University of Rhode Island
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Mercer JS, Vohr BR, McGrath MM, Padbury JF, Wallach M, Oh W. Delayed cord clamping in very preterm infants reduces the incidence of intraventricular hemorrhage and late-onset sepsis: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):1235-42. doi: 10.1542/peds.2005-1706. PMID 16585320
- [Background] Mercer JS, Vohr BR, Erickson-Owens DA, Padbury JF, Oh W. Seven-month developmental outcomes of very low birth weight infants enrolled in a randomized controlled trial of delayed versus immediate cord clamping. J Perinatol. 2010 Jan;30(1):11-6. doi: 10.1038/jp.2009.170. Epub 2009 Oct 22. PMID 19847185
- [Result] Mercer JS, Erickson-Owens DA, Vohr BR, Tucker RJ, Parker AB, Oh W, Padbury JF. Effects of Placental Transfusion on Neonatal and 18 Month Outcomes in Preterm Infants: A Randomized Controlled Trial. J Pediatr. 2016 Jan;168:50-55.e1. doi: 10.1016/j.jpeds.2015.09.068. Epub 2015 Nov 4. PMID 26547399